CLINICAL TRIAL: NCT03001895
Title: Correlation Between SUV on 18F-DCFPyL PET/CT and Gleason Score in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephan Probst, Chief of Nuclear Medicine, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-291
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL PET/CT (Experimental): 18F-DCFPyL PET/CT Scan
  Interventions: Drug: 18F-DCFPyL PET/CT

INTERVENTIONS:
Drug: 18F-DCFPyL PET/CT — 18F-DCFPyL PET/CT

SUMMARY:
Prostate specific membrane antigen (PSMA) is a unique membrane bound glycoprotein, which is overexpressed manifold on prostate cancer cells and is well-characterized as an imaging biomarker of prostate cancer. Positron emission tomography / computer tomography (PET/CT) is a nuclear medicine procedure based on the measurement of positron emission from radiolabeled tracer molecules. 18F-DCFPyL is a tracer for prostate cancer PET imaging which binds to PSMA. The strength of functional imaging methods is in distinguishing tissues according to metabolism rather than structure. Studies have shown that PET/CT imaging with 18F-DCFPyL can detect prostate cancer lesions with excellent contrast and a high detection rate even when the level of prostate specific antigen is low.

The objective of this study is to evaluate if the patient-wide SUVmax on 18F-DCFPyL PET/CT in locoregional and metastatic prostate cancer correlates with histopathologic Gleason score at initial biopsy. It is hypothesized that SUVmax will correlate positively with Gleason score. This is of interest because non-invasive risk stratification may be possible in the future.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Canada
* Male sex
* Age 18 years or older
* Previous diagnosis of prostate cancer with Gleason Score available
* ECOG performance status 0 - 3, inclusive
* Able to understand and provide written informed consent
* Under referring physician's care
* Able to tolerate the physical/logistical requirements of a PET/CT scan including lying supine for up to 40 minutes with the arms above the head and tolerating intravenous cannulation

Exclusion Criteria:

* Medically unstable patients (e.g. acute cardiac or respiratory distress or hypotensive, etc.)
* Patients who exceed the safe weight limit of the PET/CT bed (200 kg) or who cannot fit through the PET/CT bore (70 cm diameter)
* Patients with unmanageable claustrophobia

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
SUVmax on 18F-DCFPyL PET/CT | 24 hours
  Maximum standard uptake value (SUVmax) on 18F-DCFPyL PET/CT in locoregional and metastatic prostate cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No